CLINICAL TRIAL: NCT00345137
Title: Phase 1 Study of Systemic Effects of Ng-Monomethyl-L-Arginine on Renal Hemodynamics in Patients With Polycystic Kidney Disease and Chronic Glomerulonephritis
Brief Title: Effects of Systemic NO-Inhibition on Renal Hemodynamics in Patiens With Polycystic Kidney Disease and Chronic Glomerulonephritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MED.RES.HOS.1995.02.JNB
Record Dates: First submitted 2006-06-24; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2006-06

CONDITIONS: ADPKD; Glomerulonephritis
Keywords: Renal hemodynamics; Nitric oxide
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Glomerulonephritis | interventions — omega-N-Methylarginine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Ng-monomethyl-L-arginine (drug)

SUMMARY:
The study tests the hypothesis that systemic and renal nitric oxide availability is changed in polycystic kidney disease and chronic glomerulonephritis.

DETAILED DESCRIPTION:
In a randomized, placebo controlled design, the effects of systemic treatment with monomethyl-L-arginine are studied on:

1. renal hemodynamics
2. renal sodium excretion and lithium clearance
3. blood pressure and heart rate
4. plasma levels of vasoactive hormones

in patients with adult polycystic kidney disease and chronic glomerulonephrits. The results are compared with a group of healthy control subjects

ELIGIBILITY:
Inclusion Criteria:

Healthy controls

* Age 20 to 60 years
* Both men and women
* Weight below 100 kg
* Normal clinical examination and laboratory screening
* Fertile women only if using contraception
* Informed consent according to the regulations of the local etics committee

Chronic glomerulonephritis

* Biopsy veryfied chronic glomerulonephritis
* P-creatinine < 250 µmol/L
* Weight below 100 kg
* Age 20 to 60 years
* Both men and women
* Informed consent according to the regulations of the local etics committee

Adult polycystic kidney disease (APKD)

* Diagnosis of APKD by family history and renal ultrasound or renal angiography
* P-creatinine < 250 µmol/L
* Weight below 100 kg
* Age 20 to 60 years
* Both men and women
* Informed consent according to the regulations of the local etics committee

Exclusion Criteria:

Healthy controls

* History or clinical evidence of diseases of the heart and blood vessels, kidneys, liver and pancreas, endocrine organs, lungs, neoplastic disease, myocardial infarction or cerebrovascular insult as evaluated by clinical examination and laboratory screening
* Current medication
* Drugs or alcohol abuse
* Pregnancy
* Previously within one year received more than 0.2 mSV radioactive treatment or diagnostic substances
* Donation of blood less than 1 month before the experiments

Chronic glomerulonephritis

* Apart from chronic glomerulonephritis and hypertension no history of diseases of the heart and blood vessels, liver and pancreas, endocrine organs, lungs, myocardial infarction, cerebrovascular insult or neoplastic disease.
* Patients with nephrotic syndrome or secondary glomerulonephritis
* Current medication other than antihypertensive therapy
* Drugs or alcohol abuse
* Pregnancy
* Previously within one year received more than 0.2 mSV radioactive treatment or diagnostic substances

Adult polycystic kidney disease

* Apart from APKD and hypertension no history of diseases of the heart and blood vessels, liver and pancreas, endocrine organs, lungs, myocardial infarction, cerebrovascular insult or neoplastic disease.
* Current medication other than antihypertensive therapy
* Drugs or alcohol abuse
* Pregnancy
* Previously within one year received more than 0.2 mSV radioactive treatment or diagnostic substances

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Dept. of Medicine, Holstebro Hospital, 7500 Holstebro, Denmark; Jesper N Bech, MD, Ph.d., Principal Investigator — Dept. of Medicine, Holstebro Hospital, 7500 Holstebro, Denmark

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039